CLINICAL TRIAL: NCT07114965
Title: Effects Of Quadratus Lumborum Type 1 Block And Transversalis Facial Plane Block On Acute Pain In Gynecological Surgery
Acronym: GYNQLBFPB
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkay baran akkuş, specialist doctor, Ankara Diskapi Training and Research Hospital
Other Study IDs: AEŞH-EK-2025-151
Record Dates: First submitted 2025-07-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Gynecologic Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- open gynecological operations

SUMMARY:
This study was conducted to evaluate the effectiveness of Quadratus Lumborum Type 1 and Transversalis Fascial Plane blocks on postoperative acute pain in gynecology operations.

DETAILED DESCRIPTION:
In gynecological operations, especially total abdominal hysterectomy, moderate to severe postoperative pain is usually accompanied. Inadequately treated postoperative abdominal hysterectomy pain causes delayed postoperative recovery, prolonged hospital stay, chronic pain, increased chance of venous thrombosis and patient dissatisfaction. Multimodal analgesia techniques are widely used, but new evidence has shown that combinations with regional anesthesia techniques are the most effective method in postoperative pain treatment. Opioids continue to be the main step in postoperative pain treatment, despite strong evidence of their disadvantages. Opioid administration in acute postoperative pain is associated with many side effects such as sedation, pruritus, nausea and vomiting. Regional analgesia techniques used to reduce the amount of opioid used and provide effective analgesia are becoming an integral part of postoperative opioid-sparing analgesia. Open surgeries increase tissue trauma and increase inflammatory response due to high surgical stress. The reduction of pain by regional analgesia application facilitates postoperative mobilization and reduces complications. Abdominal wall blocks are performed on the principle of high-volume local anesthetic deposition within a fascial plane. Ultrasound-guided performance with continuous visualization of the needle improves placement accuracy and reduces inadvertent visceral or neurovascular injury. Abdominal wall blocks primarily provide somatic analgesia, but newer blocks can also block visceral nerves. Abdominal wall blocks provide a relatively safe alternative to epidural analgesia without the risk of motor block, hypotension, or central neuraxis. The quadratus lumborum fascial block (QLB), recently described by Blanco and modified by Sauter et al, is considered an extension of the TAP block. A local anesthetic is injected adjacent to the QL muscle, which aims to anesthetize the thoracolumbar nerves. The QL muscle is a quadrangular-shaped posterior abdominal wall muscle that inserts inferiorly on the iliac crest, cranially on the 12th rib, medially on the transverse processes of L1 to L4, and has a free lateral margin. The QL muscle is related to the PM muscle on its anterior surface and to the spinal erector muscle group on its posterior surface. The muscle is surrounded by the thoracolumbar fascia. Three techniques for QLB have been described and named according to the position of the needle tip in relation to the QL muscle: QLB type 1 or lateral; type 2 or posterior; and transmuscular, or anterior. Many case reports and randomized trials have included analgesia for gynecologic and lower abdominal surgery, Pfannenstiel incision for cesarean section, proctosigmoidectomy, hip surgery, abdominal hernioplasty, nephrectomy, and laparotomy as indications. There are several case reports with different indications for QLB for sensory block between T7 and L2. The transversalis fascial plane block is a truncal block that targets the L1 nerve branches, namely the ilioinguinal and iliohypogastric nerves. The ilioinguinal and iliohypogastric nerves originate from the lateral border of the psoas major muscle, below the 12th rib, and run along the anterior surface of the quadratus lumborum muscle. Lateral to the quadratus lumborum muscle, it initially descends deep to the transversus abdominis muscle for a variable distance and penetrates the transversus abdominis muscle to enter the transversus abdominis plane between the internal oblique and transversus abdominis muscles. This block is also an analgesic option for inguinal hernia repair, open appendectomy, and any surgical procedure involving the L1 dermatome. In this study, the investigators will evaluate the effectiveness of quadratus lumborum and transversalis fascial plane blocks, which are abdominal wall blocks, on postoperative acute pain in open gynecological operations.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* 18-80 years old women's medicines
* Open myomectomy and total abdominal hysterectomy cases

Exclusion Criteria:

* Those who do not want a block
* Patients who are allergic to local anesthetics
* Patients with coagulopathy ·
* Pregnancy
* Previous surgery in the area where the block will be applied

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gynecologic surgery
Study Population: Women who have undergone open gynecological surgery
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain between groups | day 1
  The steps of expanding the transversalis fascial plane in acute pain are being investigated against the quadratus lumborum 1 spread applied in gynecological surgery.

SECONDARY OUTCOMES:
Time to first rescue analgesic consumption | day 1
  To investigate the effects of transversalis fascial plane block versus quadratus lumborum 1 block on the recovery time and the time to first postoperative analgesic consumption in patients undergoing gynecological surgery.
total opioid consumption | day 1
  Monitoring of total opioid consumption for 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)